CLINICAL TRIAL: NCT03148067
Title: Prospective Study on the Incidence and Risk Factors for the Occurrence of Surgical Site Infection After Intramedullary Nailing of Diaphyseal Femoral and Tibial Fractures
Brief Title: Incidence and Risk Factors for Surgical Site Infection After Intramedullary Nailing of Femoral and Tibial Fractures
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Priscila Rosalba Domingos de Oliveira, MD, MSc, University of Sao Paulo
Other Study IDs: 10075
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Fracture Fixation, Intramedullary; Surgical Wound Infection
Keywords: Risk Factors; Incidence; Epidemiology
MeSH Terms: conditions — Surgical Wound Infection | interventions — Fracture Fixation, Intramedullary; Fracture Fixation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with closed or open diaphyseal femoral and tibial fractures treated through intramedullary nailing for fracture fixation
  Interventions: Procedure: Intramedullary nailing for fracture fixation

INTERVENTIONS:
Procedure: Intramedullary nailing for fracture fixation

SUMMARY:
Diaphyseal femoral and tibial fractures are in the spotlight within the traumatology-orthopedics scenario. Intramedullary nailing (IMN) remains the method of choice for treating these fractures, both open and closed ones. Occurrences of surgical site infection (SSI) related to this type of osteosynthesis are a challenge for all the professionals involved in patient healthcare. The reported incidence of SSI after IMN ranges from 0.9 to 17.5%. The majority of the data comes from retrospective studies and as part of case series descriptions, with little detail about the criteria used for defining and searching for cases of infection. Regarding the potential risk factors for this complication, previous use of external fixators, occurrence of open fractures and the severity of exposure according to the Gustilo-Anderson classification were indicated in a few retrospective studies as being possibly related to this complication. The objectives of the present observational cohort study are: 1. To determine the incidence of SSI related to IMN for fixation of diaphyseal femoral and tibial fractures in patients treated in a university traumatology and orthopedics reference hospital in São Paulo, Brazil; 2. To evaluate the risk factors related to the occurrence of this type of infection.

DETAILED DESCRIPTION:
Diaphyseal femoral and tibial fractures are a important challenge faced by the orthopedic surgeon, due to their high incidence and high social and economic impact. Currently, the observed increases in the rates of injuries secondary to traffic, work and firearms-related accidents, and also those related to sports practice, have led to significant growth of the incidence of these fractures, especially among young and economically active individuals .

Although standardized criteria for indications of conservative treatment exist, surgery is often recommended due to its better functional results and shorter rehabilitation period. Intramedullary nailing (IMN) was introduced by Küntscher in 1939 and remains the method of choice for treating these fractures, both closed and open ones, especially because the surgical technique is considered to be simple, standardized and replicable; does not cause major soft tissue damage and allows early loading. This technique is associated with a higher consolidation rate and lower incidence of complications, among which infections are included.

Surgical site infection (SSI) after internal fracture fixation is considered to be a severe, hard-to-treat complication, and it is important to remember that the presence of the implant itself favors bacterial invasion and alters local immunity, thus hampering the action of granulocytes. In addition, injury to the soft tissues adjacent to the fracture focus also hampers this immunity and favors occurrence of infections.

Although complications are less frequent than in other internal fracture fixation methods, they can occur during the postoperative period, relating to the use of IMN, and these may include SSI. Its occurrence significantly increases recovery time and treatment costs, and it compromises the long-term functional results and rehabilitation.

SSIs, including those related to IMN, are defined internationally in accordance with the criteria established in the United States (USA) by the National Healthcare Safety Network (NHSN), an agency belonging to the Centers for Disease Control and Prevention (CDC). 8 This body is responsible for healthcare-related infection surveillance actions in that country. In Brazil, as in other countries, adaptations made by the local health and epidemiological surveillance authorities are followed.

In January 2015, the NHSN made available a document with new definitions of SSI, which came into force in the USA from that moment onwards, with important changes. The period for defining infections relating to fracture fixation procedures, regardless of the type of synthesis material used, became only 90 days, instead of one year from the data of the surgery. For better evaluation, however, for the present study, the surveillance period remains one year for defining SSIs relating to IMN.

Different incidences of SSI after fixation of lower-limb fractures through IMN have been reported in the literature. Most of these have come from retrospective studies and as part of the description of series of cases of patients who underwent this procedure, with little detail about the criteria used for defining and searching for SSI cases. Only two prospective studies have so far reported the occurrence of this complication: these studies were not specifically designed for evaluating SSI and only describe its occurrence superficially, among other complications . Until recently, only Gaebler et al., in 2000, had described this complication with greater methodological rigor. In 2015, however, because of the gap in knowledge that existed, three authors published the results from retrospective studies that had been specifically designed for evaluating SSIs relating to IMN for correcting lower-limb fractures. Despite this recent interest in this subject among researchers, there continue to be no prospective studies specifically designed for investigating the incidence of this complication, or its risk factors. In Latin America, in particular, there are no studies of any kind evaluating the incidence of SSI after fixation of lower-limb fractures using IMN.

Risk factors for occurrences of surgical site infections are generally divided into those relating to the host, the surgical environment and the microbiota. For occurrences of SSI after fracture fixation procedures, the following are considered also to be risk factors: degree of energy of the associated trauma, degree of injury of the adjacent soft tissues, degree of local contamination, duration of osteosynthesis surgery and immunological status of the patient.

However, specifically with regard to risk factors relating to occurrences of SSI after fixation of lower-limb fractures through IMN, information is scarce, given that the majority of the studies that analyzed the incidence of this complication did not allow for analysis of the risk factors relating to their occurrence. Until 2015, only Gaebler et al. had published results from an analysis on these risk factors. They concluded from their retrospective study that the risk of acquiring SSI after implantation of IMNs was 22.4 times higher among patients with Gustilo III open fractures than among patients with other types of fractures. However, these authors did not evaluate the importance of other factors that are considered to be associated with occurrences of SSI after fracture fixation.

Because of the lack of information on this important subject, in 2015 three authors published results from retrospective investigations that enabled a few conclusions. Galvin et al., in their study on closed tibial fractures in American soldiers, found higher incidence of SSI after IMN in patients who presented clinical instability during the initial care, although this difference was not statistically significant.

In turn, Metsemakers et al. concluded, after an initial univariate analysis, that previous use of external fixators, occurrences of open fractures and the severity of exposure according to Gustilo-Anderson would be factors associated with occurrences of SSI, as also would greater time intervals between the fracture and its fixation through IMN. It needs to be highlighted that these authors did not define the time interval above which the risk of infection would be greater. After multiple logistic regression analysis, however, only previous external fixation remained as a factor associated with occurrence of SSI after internal fixation of the fracture with IMN. In the study conducted by Roussignol et al., only the severity of the open fracture according to the Gustilo-Anderson classification had a statistically significant correlation with occurrences of infection. Other variables, including the severity according to the AO classification, previous external fixation, and time interval between fracture and its internal fixation did not present correlations with increased incidence of SSI associated with IMN.

It needs to be emphasized that none of the studies cited that presented information on the factors associated with occurrences of SSI after fracture fixation through IMN were prospective. This shows that the medical literature still lacks information obtained using greater methodological rigor.

ELIGIBILITY:
Inclusion Criteria:

* Closed and open diaphyseal femoral and tibial fractures treated through IMN;
* Age: 16 years or older
* The patient or a person legally responsible for the patient should sign the free and informed consent statement (FICS) in order to take part in the study.

Exclusion Criteria:

* No exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were included in the research after the surgical plan for intramedullary nailing for fixation of their fractures has been defined. This inclusion could occur up to 72 hours after the surgical procedure. If a patient presented more than one diaphyseal femoral or tibial fracture that could be potentially included in the study, only the first surgically corrected fracture were considered for analysis in the study.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lucia M Lima, MD, PhD, Study Chair — Assistant Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young S, Lie SA, Hallan G, Zirkle LG, Engesaeter LB, Havelin LI. Risk factors for infection after 46,113 intramedullary nail operations in low- and middle-income countries. World J Surg. 2013 Feb;37(2):349-55. doi: 10.1007/s00268-012-1817-4. PMID 23052810
- [Background] Ozdemir B, Akesen B, Demirag B, Bilgen MS, Durak K. Long-term outcome of unreamed intramedullary nails in femur diaphyseal fractures. Ulus Travma Acil Cerrahi Derg. 2012 Mar;18(2):147-52. doi: 10.5505/tjtes.2012.19970. PMID 22792821
- [Background] Pfeifer R, Sellei R, Pape HC. The biology of intramedullary reaming. Injury. 2010 Nov;41 Suppl 2:S4-8. doi: 10.1016/S0020-1383(10)70002-4. PMID 21144926
- [Background] Petrisor B, Anderson S, Court-Brown CM. Infection after reamed intramedullary nailing of the tibia: a case series review. J Orthop Trauma. 2005 Aug;19(7):437-41. doi: 10.1097/01.bot.0000161542.93624.8d. PMID 16056073
- [Background] Ricci WM, Gallagher B, Haidukewych GJ. Intramedullary nailing of femoral shaft fractures: current concepts. J Am Acad Orthop Surg. 2009 May;17(5):296-305. doi: 10.5435/00124635-200905000-00004. PMID 19411641
- [Background] Schmidt AH, Swiontkowski MF. Pathophysiology of infections after internal fixation of fractures. J Am Acad Orthop Surg. 2000 Sep-Oct;8(5):285-91. doi: 10.5435/00124635-200009000-00002. PMID 11029556
- [Background] Horan TC, Gaynes RP. Surveillance of nosocomial infections. In:Hospital epidemiology and infection control, 3rd ed., Mayhall CG, editor. Philadelphia:Lippincott Williams & Wilkins,2004:1659-702
- [Background] Centers for Disease Control and Prevention. Surgical Site Infection (SSI) Event. Atlanta, EUA: 2016. Available in: http://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
- [Background] Court-Brown CM, Christie J, McQueen MM. Closed intramedullary tibial nailing. Its use in closed and type I open fractures. J Bone Joint Surg Br. 1990 Jul;72(4):605-11. doi: 10.1302/0301-620X.72B4.2380211.
- [Background] Alho A, Ekeland A, Stromsoe K, Folleras G, Thoresen BO. Locked intramedullary nailing for displaced tibial shaft fractures. J Bone Joint Surg Br. 1990 Sep;72(5):805-9. doi: 10.1302/0301-620X.72B5.2211761.
- [Background] Gaebler C, Berger U, Schandelmaier P, Greitbauer M, Schauwecker HH, Applegate B, Zych G, Vecsei V. Rates and odds ratios for complications in closed and open tibial fractures treated with unreamed, small diameter tibial nails: a multicenter analysis of 467 cases. J Orthop Trauma. 2001 Aug;15(6):415-23. doi: 10.1097/00005131-200108000-00006. PMID 11514768
- [Background] Galvin JW, Dannenbaum JH 4th, Tubb CC, Poepping TP, Grassbaugh JA, Arrington ED. Infection Rate of Intramedullary Nailing in Closed Fractures of the Femoral Diaphysis After Temporizing External Fixation in an Austere Environment. J Orthop Trauma. 2015 Sep;29(9):e316-20. doi: 10.1097/BOT.0000000000000327. PMID 25785355
- [Background] Metsemakers WJ, Handojo K, Reynders P, Sermon A, Vanderschot P, Nijs S. Individual risk factors for deep infection and compromised fracture healing after intramedullary nailing of tibial shaft fractures: a single centre experience of 480 patients. Injury. 2015 Apr;46(4):740-5. doi: 10.1016/j.injury.2014.12.018. Epub 2014 Dec 27. PMID 25583638
- [Background] Roussignol X, Sigonney G, Potage D, Etienne M, Duparc F, Dujardin F. Secondary nailing after external fixation for tibial shaft fracture: risk factors for union and infection. A 55 case series. Orthop Traumatol Surg Res. 2015 Feb;101(1):89-92. doi: 10.1016/j.otsr.2014.10.017. Epub 2015 Jan 13. PMID 25595427
- [Background] Winquist RA, Hansen ST Jr, Clawson DK. Closed intramedullary nailing of femoral fractures. A report of five hundred and twenty cases. J Bone Joint Surg Am. 1984 Apr;66(4):529-39. PMID 6707031
- [Background] Court-Brown CM, McQueen MM, Quaba AA, Christie J. Locked intramedullary nailing of open tibial fractures. J Bone Joint Surg Br. 1991 Nov;73(6):959-64. doi: 10.1302/0301-620X.73B6.1955445.
- [Background] Court-Brown CM, Keating JF, McQueen MM. Infection after intramedullary nailing of the tibia. Incidence and protocol for management. J Bone Joint Surg Br. 1992 Sep;74(5):770-4. doi: 10.1302/0301-620X.74B5.1527132.
- [Background] Keating JF, Blachut PA, O'Brien PJ, Court-Brown CM. Reamed nailing of Gustilo grade-IIIB tibial fractures. J Bone Joint Surg Br. 2000 Nov;82(8):1113-6. doi: 10.1302/0301-620x.82b8.10566. PMID 11132268
- [Background] Court-Brown CM. Reamed intramedullary tibial nailing: an overview and analysis of 1106 cases. J Orthop Trauma. 2004 Feb;18(2):96-101. doi: 10.1097/00005131-200402000-00007. No abstract available. PMID 14743029
- [Background] Halvorson JJ, Barnett M, Jackson B, Birkedal JP. Risk of septic knee following retrograde intramedullary nailing of open and closed femur fractures. J Orthop Surg Res. 2012 Feb 17;7:7. doi: 10.1186/1749-799X-7-7. PMID 22340770
- [Background] Sie E, Kacou A, Traore A, Sery B, Lambin Y. Primary unreamed and unlocked intramedullary nailing of femoral shaft fractures. Malays Orthop J. 2012 Nov;6(3):13-7. doi: 10.5704/MOJ.1207.014. PMID 25279049
- [Background] Salem KH. Unreamed intramedullary nailing in distal tibial fractures. Int Orthop. 2013 Oct;37(10):2009-15. doi: 10.1007/s00264-013-1998-y. Epub 2013 Jul 28. PMID 23892464
- [Background] AO Foundation. AO/OTA Fracture and dislocation classification. Davos, Suíça: 2014. Available in: https://www.aofoundation.org/Structure/resource/AO-OTA-Fracture-Dislocation-Classification/Pages/AO-OTA-Fracture-Dislocation-Classification-Long-Bones.aspx
- [Background] Gustilo RB, Anderson JT. Prevention of infection in the treatment of one thousand and twenty-five open fractures of long bones: retrospective and prospective analyses. J Bone Joint Surg Am. 1976 Jun;58(4):453-8. PMID 773941
- [Background] Gustilo RB, Mendoza RM, Williams DN. Problems in the management of type III (severe) open fractures: a new classification of type III open fractures. J Trauma. 1984 Aug;24(8):742-6. doi: 10.1097/00005373-198408000-00009. PMID 6471139
- [Background] Maragakis LL, Perl TM. Basics of surgical site infection surveillance and prevention. In: Practical Healthcare Epidemiology, 3rd ed., Lautenbach E, Woeltje KF, Malani PN, editor. Chicago: The University of Chicago Press, 2010:173-185
- [Background] Oliveira PR, Carvalho VC, da Silva Felix C, de Paula AP, Santos-Silva J, Lima AL. The incidence and microbiological profile of surgical site infections following internal fixation of closed and open fractures. Rev Bras Ortop. 2016 Feb 2;51(4):396-9. doi: 10.1016/j.rboe.2015.09.012. eCollection 2016 Jul-Aug. PMID 27517016
- [Background] Silva AGP, Silva FBA, Godoy-Santos AL, Luzo CAM, Sakaki MH, Zumiotti AV. Infecção pós-estabilização intramedular das fraturas diafisárias dos membros inferiores: Protocolo de tratamento. Acta Ortop Bras 2008;16:266-9

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients: 221 Patients with closed or open diaphyseal femoral and tibial fractures treated through intramedullary nailing for fracture fixation were included and completed follow up
  Intramedullary nailing for fracture fixation
Period: Overall Study
Arm/Group | Patients
Started | 225
Completed | 221
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 221 patients were included and completed follow up
Groups:
- Patients: Patients with closed or open diaphyseal femoral and tibial fractures treated through intramedullary nailing for fracture fixation
  Intramedullary nailing for fracture fixation
Arm/Group | Patients
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 173
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 221

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Surgical Site Infection (SSI) Relating to Intramedullary Nailing for Fixation of Diaphyseal Femoral and Tibial Fractures
Description: Patients who present signs of infection in the region of the surgery under evaluation or who describe alterations compatible with SSI, or whose records mention signs or symptoms compatible with the definitions of SSI, are considered to be cases with evolution to infection. Patients included in the study who, during routine or emergency care present a condition (according to the researchers' evaluation) suggestive of a SSI associated with intramedullary nailing are considered to be cases of infection
Time Frame: one year after surgery
Population: 221 patients included in the study completed the planned follow up period. In total, 26 cases of infection were observed, with an incidence of 11.8%.
Measure: Count of Participants; unit: Participants
Groups:
- Patients: 221 Patients with closed or open diaphyseal femoral and tibial fractures treated through intramedullary nailing for fracture fixation were included and completed follow up. In total, 26 cases of infection were observed after 12 months of follow-up, with an incidence of 11.8%.
Arm/Group | Patients
Number analyzed (Participants) | 221
Participants
  Patients with infection | 26
  Patients without infection | 195

2. Secondary Outcome: Possible Risk Factors Related to Occurrence of SSI After Intramedullary Nailing
Description: Patient-related factors: age; gender; body mass index; duration of preoperative hospitalization; infection in other foci; presence of immunosuppressive conditions; physical status classification according to ASA; occurrences of multiple trauma and ISS score; injury etiology; exposure time (for open fractures); AO fracture classification; soft-tissue injury classification; Gustilo-Anderson open fracture classification; stay at other hospital before transference; use of external fixation; previous surgical manipulation and use of blood products. Factors relating to the surgery: wound classification according to potential for contamination; surgery length; hair removal; antibiotic prophylaxis or therapy; use of drains; patient temperature and oxygenation; type of nail used (anterograde or retrograde); reaming; primary closure; necessity for a skin-muscle flap and use of negative-pressure wound therapy. Microbiota-related factors: evaluation of colonization by S. aureus and A. baumannii.
Time Frame: one year after surgery
Population: Previous use of external fixations (OR 2.53) and need for soft tissue reconstruction (OR 10.94) were associated to surgical site infections after intramedular nailing
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Patients
Number analyzed (Participants) | 221
odds ratio
  Previous use of external fixation | 2.53 [0.98 to 6.56]
  Need for soft tissue reconstruction | 10.94 [3.07 to 38.92]

ADVERSE EVENTS:
Time Frame: 18 months
Description: 26 cases of infection were observed after 12 months of follow-up. One patient died from infection.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 1/221
Serious Adverse Events (participants affected / at risk) | 26/221
Other Adverse Events (participants affected / at risk) | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=221)
Surgical site infection (Infections and infestations) | 26 (26)

LIMITATIONS AND CAVEATS:
Hyperglicemia was not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03148067/Prot_SAP_000.pdf